CLINICAL TRIAL: NCT06193057
Title: Comparison of Customized and Standard Total Ankle Prostheses: a Pilot Study
Brief Title: Comparison of Customized and Standard Total Ankle Prostheses
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istituto Ortopedico Rizzoli (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 3POD-TAR
Record Dates: First submitted 2023-12-21; First posted 2024-01-05 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Ankle Osteoarthritis
Keywords: replacement; customized; TAR; arthroplasty; radiographic angles; clinical scores
MeSH Terms: interventions — Arthroplasty, Replacement, Ankle

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Traditional (Active Comparator): In the STANDARD group, patients will undergo a primary TAR by implanting a prosthetic model of a standard design, that is the same for all using the usual surgical technique and instrumentation (based on the use of external leg guidance)
  Interventions: Procedure: Total ankle arthroplasty
- Custom (Experimental): In the PERSONALIZED group, patients will undergo a primary TAR by implanting a prosthetic model with a design specifically based on each patient's actual ankle morphology and using PSI surgical technique and instrumentation.
  Interventions: Procedure: Total ankle arthroplasty

INTERVENTIONS:
Procedure: Total ankle arthroplasty — Patients who underwent ankle prosthesis implantation procedure with an anterior approach were involved in a longitudinal skin incision of about 12-15cm anterior to the tibio-tarsal joint in supine position. Once the deep layers were reached, passing through the anterior tibial tendon and extensor hallucis longus tendon sheath, the tibio-tarsal joint was then exposed. The operator proceeds to astragalic and tibial resections, once the appropriate size of implants was selected, the final components were implanted. In both groups, the basic prosthetic design approach will be 'three-component,' that is, with congruent mobile meniscus interposed between the tibial and astragalic components. At the end of the procedure, orthopedic walker boot was placed for 3 weeks, and progressive weight allowed.
  Other Names: Total ankle arthroplasty with anterior approach

SUMMARY:
The objective of this study is to compare primary total ankle replacement (TAR) performed with a customized procedure (prostheses customized for each patient based on his or her ankle morphology reconstructed from tomographic scans, and implanted via cutting guides customized for the patient) with standard primary TARs, considering: objective radiological results, subjective patient outcomes, and overall costs of both procedures

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects older than 40 years and younger than 75 years (≥ 40 age ≤ 75 years) with arthrosis at the unilateral tibio-tarsal joint who are candidates for primary total ankle replacement.
* Consenting patients and able to complete scheduled study procedures and follow-up evaluations.
* Patients who have signed the "informed consent" approved by the Ethics Committee.

Exclusion Criteria:

* Social conditions (homeless patients, with restrictions on personal freedom)
* ASA 3 and 4
* Deep venous insufficiency Lower limbs
* History of Erisipelas lower limbs
* Neurological or psychocognitive disorders
* neurological diseases
* Axial deformities of ankle >15°
* Personal or family history of DVT or EP
* Prosthetic and/or arthrodesis surgeries at another lower extremity joint except that candidate for ankle prosthesis)
* Pregnant women
* Patients with rheumatic diseases
* Patients that requires ancillary surgical procedures

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2023-07-26 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2027-04-26 (Estimated)

PRIMARY OUTCOMES:
Ankle radiographic angles | at baseline (day 0)
  Patients will be evaluated by how many degrees the postoperative ankle angle in loading, either varo-valgus (frontal alignment) or dorsi-plantar differs from the corresponding physiological angles (4° and 0°, respectively) when implanting a customized primary TAR (PERSONALIZED group) versus a standard primary TAR (STANDARD group) according to normal surgical practice.
Ankle radiographic angles | 3 months
  Patients will be evaluated by how many degrees the postoperative ankle angle in loading, either varo-valgus (frontal alignment) or dorsi-plantar differs from the corresponding physiological angles (4° and 0°, respectively) when implanting a customized primary TAR (PERSONALIZED group) versus a standard primary TAR (STANDARD group) according to normal surgical practice.
Ankle radiographic angles | 6 months
  Patients will be evaluated by how many degrees the postoperative ankle angle in loading, either varo-valgus (frontal alignment) or dorsi-plantar differs from the corresponding physiological angles (4° and 0°, respectively) when implanting a customized primary TAR (PERSONALIZED group) versus a standard primary TAR (STANDARD group) according to normal surgical practice.
Ankle radiographic angles | 12 months
  Patients will be evaluated by how many degrees the postoperative ankle angle in loading, either varo-valgus (frontal alignment) or dorsi-plantar differs from the corresponding physiological angles (4° and 0°, respectively) when implanting a customized primary TAR (PERSONALIZED group) versus a standard primary TAR (STANDARD group) according to normal surgical practice.
Ankle radiographic angles | 18 months
  Patients will be evaluated by how many degrees the postoperative ankle angle in loading, either varo-valgus (frontal alignment) or dorsi-plantar differs from the corresponding physiological angles (4° and 0°, respectively) when implanting a customized primary TAR (PERSONALIZED group) versus a standard primary TAR (STANDARD group) according to normal surgical practice.

SECONDARY OUTCOMES:
Short form 12 | at baseline (day 0)
  The SF-12 health questionnaire is a generic standardized instrument for fast, economic and disease-border acquisition of health-related quality of life."
Short form 12 | 3 months
  The SF-12 health questionnaire is a generic standardized instrument for fast, economic and disease-border acquisition of health-related quality of life."
Short form 12 | 6 months
  The SF-12 health questionnaire is a generic standardized instrument for fast, economic and disease-border acquisition of health-related quality of life."
Short form 12 | 12 months
  The SF-12 health questionnaire is a generic standardized instrument for fast, economic and disease-border acquisition of health-related quality of life."
Short form 12 | 18 months
  The SF-12 health questionnaire is a generic standardized instrument for fast, economic and disease-border acquisition of health-related quality of life."
Visual Analogic Scale | at baseline (day 0)
  Visual Analogue Scale (VAS) is a measurement instrument that measures a characteristic or attitude that is believed to range across a continuum of values and cannot easily be directly measured; operationally a VAS is usually a horizontal line, 100 mm in length, anchored by word descriptors at each end, where the patient marks on the line the point that they feel represents their perception of their current state. The VAS score is determined then by measuring in millimetres from the left hand end of the line to the point that the patient marks.
Visual Analogic Scale | 3 months
  Visual Analogue Scale (VAS) is a measurement instrument that measures a characteristic or attitude that is believed to range across a continuum of values and cannot easily be directly measured; operationally a VAS is usually a horizontal line, 100 mm in length, anchored by word descriptors at each end, where the patient marks on the line the point that they feel represents their perception of their current state. The VAS score is determined then by measuring in millimetres from the left hand end of the line to the point that the patient marks.
Visual Analogic Scale | 6 months
  Visual Analogue Scale (VAS) is a measurement instrument that measures a characteristic or attitude that is believed to range across a continuum of values and cannot easily be directly measured; operationally a VAS is usually a horizontal line, 100 mm in length, anchored by word descriptors at each end, where the patient marks on the line the point that they feel represents their perception of their current state. The VAS score is determined then by measuring in millimetres from the left hand end of the line to the point that the patient marks.
Visual Analogic Scale | 12 months
  Visual Analogue Scale (VAS) is a measurement instrument that measures a characteristic or attitude that is believed to range across a continuum of values and cannot easily be directly measured; operationally a VAS is usually a horizontal line, 100 mm in length, anchored by word descriptors at each end, where the patient marks on the line the point that they feel represents their perception of their current state. The VAS score is determined then by measuring in millimetres from the left hand end of the line to the point that the patient marks.
Visual Analogic Scale | 18 months
  Visual Analogue Scale (VAS) is a measurement instrument that measures a characteristic or attitude that is believed to range across a continuum of values and cannot easily be directly measured; operationally a VAS is usually a horizontal line, 100 mm in length, anchored by word descriptors at each end, where the patient marks on the line the point that they feel represents their perception of their current state. The VAS score is determined then by measuring in millimetres from the left hand end of the line to the point that the patient marks.
American Orthopedic Foot and Ankle Score | at baseline (day 0)
  This Score, based on a questionnaire, consists of points given to nine items divided in three categories: pain (40 points), functional aspects (50 points) and alignment (10 points) totaling 100 points, the extreme which represent a normal foot and ankle complex.
American Orthopedic Foot and Ankle Score | 3 months
  The AOFAS, based on a questionnaire, consists of points given to nine items divided in three categories: pain (40 points), functional aspects (50 points) and alignment (10 points) totaling 100 points, the extreme which represent a normal foot and ankle complex.
American Orthopedic Foot and Ankle Score | 6 months
  The AOFAS, based on a questionnaire, consists of points given to nine items divided in three categories: pain (40 points), functional aspects (50 points) and alignment (10 points) totaling 100 points, the extreme which represent a normal foot and ankle complex.
American Orthopedic Foot and Ankle Score | 12 months
  The AOFAS, based on a questionnaire, consists of points given to nine items divided in three categories: pain (40 points), functional aspects (50 points) and alignment (10 points) totaling 100 points, the extreme which represent a normal foot and ankle complex.
American Orthopedic Foot and Ankle Score | 18 months
  The AOFAS, based on a questionnaire, consists of points given to nine items divided in three categories: pain (40 points), functional aspects (50 points) and alignment (10 points) totaling 100 points, the extreme which represent a normal foot and ankle complex.
Ankle Range of motion | at baseline (day 0)
  Degrees of active and passive joint excursion of the ankle in dorsiflexion and plantarflexion. Normal ankle dorsiflexion is about 20°-30°, while normal plantarflexion is about 30°-50°.
Ankle Range of motion | 3 months
  Degrees of active and passive joint excursion of the ankle in dorsiflexion and plantarflexion. Normal ankle dorsiflexion is about 20°-30°, while normal plantarflexion is about 30°-50°.
Ankle Range of motion | 6 months
  Degrees of active and passive joint excursion of the ankle in dorsiflexion and plantarflexion. Normal ankle dorsiflexion is about 20°-30°, while normal plantarflexion is about 30°-50°.
Ankle Range of motion | 12 months
  Degrees of active and passive joint excursion of the ankle in dorsiflexion and plantarflexion. Normal ankle dorsiflexion is about 20°-30°, while normal plantarflexion is about 30°-50°.
Ankle Range of motion | 18 months
  Degrees of active and passive joint excursion of the ankle in dorsiflexion and plantarflexion. Normal ankle dorsiflexion is about 20°-30°, while normal plantarflexion is about 30°-50°.

CONTACTS AND LOCATIONS:
Locations (1):
- Rizzoli Orthopaedic Institute, Bologna, BO, Italy

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Result] Shane A, Sahli H. Total Ankle Replacement Options. Clin Podiatr Med Surg. 2019 Oct;36(4):597-607. doi: 10.1016/j.cpm.2019.06.005. PMID 31466570
- [Result] Foran IM, Vafek EC, Bohl DD, Lee S, Hamid KS. Quality Assessment of Modern Total Ankle Arthroplasty Clinical Outcomes Research. J Foot Ankle Surg. 2022 Jan-Feb;61(1):7-11. doi: 10.1053/j.jfas.2021.05.011. Epub 2021 Jun 10. PMID 34244049
- [Result] Mosca M, Caravelli S, Vocale E, Massimi S, Censoni D, Di Ponte M, Fuiano M, Zaffagnini S. Clinical Radiographical Outcomes and Complications after a Brand-New Total Ankle Replacement Design through an Anterior Approach: A Retrospective at a Short-Term Follow Up. J Clin Med. 2021 May 23;10(11):2258. doi: 10.3390/jcm10112258. PMID 34071032
- [Result] Malerba F, Benedetti MG, Usuelli FG, Milani R, Berti L, Champlon C, Leardini A. Functional and clinical assessment of two ankle arthrodesis techniques. J Foot Ankle Surg. 2015 May-Jun;54(3):399-405. doi: 10.1053/j.jfas.2014.09.007. Epub 2014 Nov 26. PMID 25434867
- [Result] Goldberg AJ, Chowdhury K, Bordea E, Hauptmannova I, Blackstone J, Brooking D, Deane EL, Bendall S, Bing A, Blundell C, Dhar S, Molloy A, Milner S, Karski M, Hepple S, Siddique M, Loveday DT, Mishra V, Cooke P, Halliwell P, Townshend D, Skene SS, Dore CJ; TARVA Study Group; Brown R, Butler M, Chadwick C, Clough T, Cullen N, Davies M, Davies H, Harries B, Khoo M, Makwana N, Murty A, Najefi A, O'Donnell P, Raglan M, Thomas R, Torres P, Welck M, Winson I, Zaidi R. Total Ankle Replacement Versus Arthrodesis for End-Stage Ankle Osteoarthritis: A Randomized Controlled Trial. Ann Intern Med. 2022 Dec;175(12):1648-1657. doi: 10.7326/M22-2058. Epub 2022 Nov 15. PMID 36375147
- [Result] Belvedere C, Siegler S, Fortunato A, Caravaggi P, Liverani E, Durante S, Ensini A, Konow T, Leardini A. New comprehensive procedure for custom-made total ankle replacements: Medical imaging, joint modeling, prosthesis design, and 3D printing. J Orthop Res. 2019 Mar;37(3):760-768. doi: 10.1002/jor.24198. Epub 2019 Jan 3. PMID 30537247
- [Result] Faldini C, Mazzotti A, Belvedere C, Durastanti G, Panciera A, Geraci G, Leardini A. A new ligament-compatible patient-specific 3D-printed implant and instrumentation for total ankle arthroplasty: from biomechanical studies to clinical cases. J Orthop Traumatol. 2020 Sep 2;21(1):16. doi: 10.1186/s10195-020-00555-7. PMID 32876778
- [Result] Mazzotti A, Arceri A, Zielli S, Bonelli S, Viglione V, Faldini C. Patient-specific instrumentation in total ankle arthroplasty. World J Orthop. 2022 Mar 18;13(3):230-237. doi: 10.5312/wjo.v13.i3.230. eCollection 2022 Mar 18. PMID 35317257
- [Result] Brinkmann EJ, Fitz W. Custom total knee: understanding the indication and process. Arch Orthop Trauma Surg. 2021 Dec;141(12):2205-2216. doi: 10.1007/s00402-021-04172-9. Epub 2021 Oct 15. PMID 34652517
- [Result] Leardini A, Belvedere C, de Cesar Netto C. Total Ankle Replacement: Biomechanics of the Designs, Clinical Outcomes, and Remaining Issues. Foot Ankle Clin. 2023 Mar;28(1S):e1-e14. doi: 10.1016/j.fcl.2023.01.001. Epub 2023 Mar 1. PMID 36935170
- [Result] Ferraro D, Siegler S, Belvedere C, Ruiz M, Leardini A. Effect of artificial surface shapes and their malpositioning on the mechanics of the replaced ankle joint for possible better prosthesis designs. Clin Biomech (Bristol). 2021 Dec;90:105489. doi: 10.1016/j.clinbiomech.2021.105489. Epub 2021 Sep 17. PMID 34560346
- [Result] Pavani C, Belvedere C, Ortolani M, Girolami M, Durante S, Berti L, Leardini A. 3D measurement techniques for the hindfoot alignment angle from weight-bearing CT in a clinical population. Sci Rep. 2022 Oct 7;12(1):16900. doi: 10.1038/s41598-022-21440-9. PMID 36207422
- [Result] Kitaoka HB, Alexander IJ, Adelaar RS, Nunley JA, Myerson MS, Sanders M. Clinical rating systems for the ankle-hindfoot, midfoot, hallux, and lesser toes. Foot Ankle Int. 1994 Jul;15(7):349-53. doi: 10.1177/107110079401500701. PMID 7951968
- [Result] Boeckstyns MEH, Backer M. Reliability and validity of the evaluation of pain in patients with total knee replacement. Pain. 1989 Jul;38(1):29-33. doi: 10.1016/0304-3959(89)90069-9. PMID 2780060
- [Result] Hagell P, Westergren A, Arestedt K. Beware of the origin of numbers: Standard scoring of the SF-12 and SF-36 summary measures distorts measurement and score interpretations. Res Nurs Health. 2017 Aug;40(4):378-386. doi: 10.1002/nur.21806. PMID 28732149